CLINICAL TRIAL: NCT04957628
Title: Implementation of Tailored Interventions to Treat Harmful Alcohol and Drug Use for Medical Patients in Norwegian Hospitals and the Municipality Service - AlcoTail
Brief Title: AlcoTail - Implementation of Tailored Interventions
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Lovisenberg Diakonale Hospital (Other); Oslo Municipality (Other Government)
Responsible Party: Principal Investigator, Stig Tore Bogstrand, Head of Research, Oslo University Hospital
Other Study IDs: 31052
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Consumption; Psychoactive Substance Use
Keywords: Alcohol; Psychoactive drugs; Intervention; Somatic patients
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Left-over material (EDTA full blood) from routine diagnostic purposes will be collected from all study participants once they are enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 2500 participants will be recruited before the intervention procedures are implemented at the respective hospitals. Baseline data on alcohol, psychoactive medicinal and illicit drug use (AUDIT-4 and DUDIT), stages-of-change questionnaire on alcohol, medicinal drugs and illicit drug use, and mental distress will be recorded. Left-over full blood from routine diagnostic testing will be collected and analyzed for alcohol biomarkers (ethanol and phosphatidylethanol (PEth)) and psychoactive medicinal and illicit drugs. The participants in the control group will receive acute medical treatment according to hospital procedures. After 12 months, the data from baseline will be coupled to data from patient journals and data from relevant registries.
- Case group: 2500 participants will be recruited after the intervention procedures are implemented. Baseline data on alcohol, psychoactive medicinal and illicit drug use, stages-of-change questionnaires, and mental distress will be recorded. Left-over blood from diagnostic testing will be collected and analyzed for alcohol biomarkers (ethanol and phosphatidylethanol (PEth)) and psychoactive medicinal and illicit drugs. The participants in the case group will receive treatment according to new hospital procedures, including screening for harmful alcohol use and non-prescribed use of psychoactive medicinal drugs and intervention. If feasible, a new blood sample will be collected 2 months after inclusion, which will be analyzed for PEth. After 12 months, the data from baseline will be coupled to patient journals and relevant registries.
  Interventions: Behavioral: Harmful alcohol use treatment; Behavioral: Non-prescribed psychoactive medicinal use treatment

INTERVENTIONS:
Behavioral: Harmful alcohol use treatment — Patients identified through routine hospital screening as having a potentially harmful alcohol use (AUDIT-C 4-6 points (men) / 3-5 points (women) will receive information about the possible harmful effects of their drinking and will be advised to reduce their consumption. Patients identified with more excessive drinking patterns (AUDIT-C > 6 (men) / > 5 (women) will be assessed with blood sample analysis of relevant alcohol biomarkers, psychological assessments for alcohol addiction and withdrawal symptoms, and if necessary referral to alcohol addiction treatment. Patients with severe withdrawal symptoms will be put in CIWA-Ar observation.
  Groups: Case group
Behavioral: Non-prescribed psychoactive medicinal use treatment — Patients with prescription on psychoactive medicinal drugs are pharmacologically assessed using serum sample analysis. Patients identified with discrepancy in prescribed doses and serum concentrations will have doses adjusted, or be referred to addiction treatment. Patients identified with psychoactive medicinal drugs other than those prescribed will be advised to quit those medications, or be referred to addiction treatment.
  Groups: Case group

SUMMARY:
This study aims to investigate the implementation and real-world effects of an intervention for harmful use of alcohol and psychoactive medicinal drugs among hospital inpatients. Due to the negative impact of alcohol consumption on health outcomes, a call for action has been made by the Norwegian Ministry of Health, with focus on screening patients for alcohol consumption and evidence-based tailored interventions for those with medium or high consumption. In addition, non-prescribed use of psychoactive medicinal drugs, or concomitant use with alcohol, can also have negative health effects, therefore improved monitoring of the use of these are warranted. Interventions will be introduced as routine procedures at Norwegian hospitals in the upcoming year, and 2500 patients receiving acute medical care will be included in the control group before the intervention is implemented, and 2500 patients in the case group after the implementation is effectuated. This study will evaluate the implementation process using baseline data on self-reported alcohol- and psychoactive medicine use, motivation to reduce consumption and mental distress. In addition, left-over blood samples used for diagnostic purposes will be collected and analyzed for alcohol, psychoactive medicinal and illicit drugs. After 12 months baseline data will be coupled to patient journal data and relevant registry data in order to evaluate the effects of the intervention.

DETAILED DESCRIPTION:
Patients included in the study before the implementation of the intervention protocols will be assigned to the control group. These patients will receive acute medical care according to current procedures. Patients included in the study after implementation of intervention protocols will be assigned to the case group. In addition to acute medical care, these patients will be routinely screened for harmful alcohol consumption using Alcohol Use Disorder Identification Test (AUDIT-C). Patients scoring < 4 points (men) / 3 points (women) will not receive any intervention. Patients scoring 4-6 points (men) / 3-5 points (women) will be informed about the possible harmful effects of their consumption and will be advised to reduce their consumption. From patients scoring > 6 points (men) >5 points (women) a blood sample will be collected and analyzed for relevant biomarkers. They will be further evaluated using Prediction of Alcohol Withdrawal Severity Scale (PAWSS). Patients at risk of developing delirium tremens will be treated according to Clinical Institute Withdrawal Assessment (CIWA-Ar) procedures, and referred to specialized alcohol addiction treatment. Patients in the case group that has prescription(s) for psychoactive medicinal drugs will also be routinely evaluated by pharmacological assessment of drug concentration in serum samples. If there is a discrepancy between prescribed dose and serum concentration, or medicinal drugs other than those being prescribed are found, the patient will be advised to use medicines according to prescription or have their prescribed dosage altered. If necessary, the patient will be referred to specialized drug addiction treatment.

The patients will be recruited from 3 hospitals: Oslo University Hospital, Lovisenberg Diakonale Hospital (Oslo) and St Olav Hospital (Trondheim). The recruitment period will be approximately 4 months for the control group and 4 months for the case group, and estimations based on previous admission numbers for the 3 hospitals results in about 2500 patients in each group.

For the study, research personnel will approach the eligible patients once they have been admitted to various medical wards. The personnel will give the patients written and verbal information about the study, and the patients who agree to be part of the study will sign a written consent. Baseline data will be recorded for all patients included in the control and case groups. These data include:

* Alcohol use past 12 months, Alcohol Use Disorder Identification Test (AUDIT-4)
* Alcohol use last 24 hours,
* Stages-of-change questionnaire on alcohol, psychoactive medicinal and/or illicit drug use past 12 months,
* Non-prescribed use of psychoactive medicinal drugs past 12 months
* Drug Use Disorder Identification Test (DUDIT)
* Stages-of-change questionnaire on psychoactive medicinal drugs or illicit drugs
* Symptoms Checklist (SCL-5)
* Left-over blood samples used for routine diagnostic testing will be collected and analyzed for ethanol, phosphatidylethanol (PEth; biomarker for alcohol use last 3 weeks), diazepam, N-desmethyldiazepam, clonazepam, oxazepam, nitrazepam, alprazolam, zopiclone, zolpidem, morphine, codeine, oxycodone, buprenorphine, methadone, tramadol, amphetamine, methamphetamine, ecstasy (MDMA), THC, cocaine and benzoylecgonine.
* Patients in the case group will be invited to submit a new blood sample for PEth analysis 2 months after inclusion.
* After 12 months, baseline data will be coupled to the following data from the patient journal: date and time of admission, days and hours spent at bed-post and intensive care, number of previous hospital admissions, ICD-10 diagnoses at discharge, level of care, AUDIT-C score, ethanol and PEth concentration in blood, psychoactive medicine concentration in serum, CIWA-Ar, Glasgow Coma Scale (GCS) score, first triage at hospital, medicinal curve at admission, marital status, employment status, care status for children under 18 years of age. Data will also be coupled to various registry data; The Norwegian Patient Registry: number of admissions in the specialist health care service 5 years prior to admission, number of treatments with main diagnosis from ICD-10 the within 5 years prior to admission, number of admissions to interdisciplinary specialist treatment within 5 years after admission, number of admissions within 5 years after admission; The Social Security Database: performance status at time of admission and 1 year after; The Norway Control and Payment of Health Reimbursement (KUHR) Database and the Norwegian Registry for Primary Health Care: patients use of institutions and other primary health care services such as home nursing and nursing homes 5 years prior to and 5 years after admission, overview of drug use diagnoses; the Norwegian Prescription Registry: medication prescribed 5 years prior to and 5 years after admission; and the Cause of Death Registry: cause of death within 5 years after admission.

The database from baseline (questionnaires and blood sample analysis), patient journal data and the various registry data collected from each included patient will be treated de-identified. The questionnaires will be in an online-format ("Nettskjema"), and the data will be submitted directly in a secure database provided by the University of Oslo, called Services for Sensitive Data (short form "TSD" in Norwegian).

In the final database, missing values in variables will result in exclusion of that patient in statistical analysis (when the variable with missing value is part of a specific analysis). Statistical analyses will include:

For the alcohol intervention:

* To control for baseline measures, multiple models for repeated measures will be used to evaluate anticipated differences between the intervention and the control groups. For the continuous outcomes (number of admissions and GP visits) linear mixed models will be fitted, for binary outcomes models with log link or Poisson link function will be used.

For the psychoactive medicinal drug intervention:

* Multiple mixed effects models for repeated measures will be fitted. The three different institutions will be entered as random effects, while selected covariates as patients' age and gender will be modeled as fixed effects. Continuous outcomes (serum concentrations) will be analyzed using linear mixed models, while changes in prescriptions with the outcome being binary will be modeled using mixed models with log or Poission link function. The results will be expressed as effect sizes (for linear models) or relative risks (RR) for models of binary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Medical wards

Exclusion Criteria:

* Inability to understand written and verbal Norwegian
* Cognitive or mental inability to consent to participation
* Injury or planned surgery as primary reason for admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to medical wards at Oslo University Hospital, Lovisenberg Diakonale Hospital and St Olav Hospital during recruitment periods that are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in alcohol consumption | 2 months
  Assess changes in alcohol consumption for patients identified with medium or high alcohol consumption will be assessed using the blood biomarker phosphatidyletanol (PEth), measured in nM. PEth will be measured at baseline and after 2 months, if feasible.
Changes in use of psychoactive medicinal drugs | 12 months
  Assess changes in use of psychoactive substances, if the patient is adviced to reduce. Measured in changes in prescription from the prescription database. Measuerd in defined daily dose (DDD).

SECONDARY OUTCOMES:
Changes in patient's health outcomes | 12 months
  Assess changes in patient's health outcomes defined as changes in diagnostic parameters in health registries, measured by changes in registered ICD-10 codes.
Changes in patient's use of health care services | 12 months
  Assess changes in use of secondary health care services, measured by number of hospital admissions,
Changes in patient's referals to specialist health care | 12 months
  Assess changes in referrals to specialist health care, measured by number of referals.
Changes in patient's use of primary healthcare | 12 months
  Assess changes in use of primary health care measured by number of PCP visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No